CLINICAL TRIAL: NCT05438498
Title: Real World Evaluation of the Effectiveness of AZD7442 for Prevention of SARS-CoV-2 Infection in Immuno-Suppressed Cancer Patients
Brief Title: Real World Evaluation of the Effectiveness of AZD7442 for Prevention of SARS-CoV-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA withdrew EUA for AZD7442
Sponsor: MediMergent, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ESR 22-21698
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: SARS-CoV-2 Infection
Keywords: solid tumor; hematologic malignancy
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Intervention Model Description: multi-center, prospective, open-label, pragmatic evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evusheld (AZD7442) (Other): Evusheld (tixagevimab+cilgavimab) 600 mg IM or IV administered one time only
  Interventions: Drug: Evusheld (tixagevimab+cilgavimab) IM or IV

INTERVENTIONS:
Drug: Evusheld (tixagevimab+cilgavimab) IM or IV — Evusheld (tixagevimab 300 mg +cilgavimab 300 mg) IM or IV
  Other Names: AZD7442

SUMMARY:
If a treated cancer patient cannot make antibodies to a Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Emergency Use Authorization (EUA) or approved vaccine, their risk for infection and its sequelae are significantly increased. The Astra-Zeneca Immuno-Suppressed Program (AISP) is designed to address whether a patient treated for cancer who receives a single-dose of Evusheld (AZD7442) 600 mg IM or IV will maintain a stable/protective effect against symptomatic SARS-CoV-2 infection including SARS-CoV-2 related hospitalization and/or SARS-CoV-2 related death up to 12 months post-baseline. The program will focus on patients with cancer who have been treated with chemotherapy, immunotherapy, targeted therapy, other therapy or combination therapy with or without radiation therapy within 12 months prior to enrollment, are willing/able to receive one IM or IV injection of Evusheld, are able to complete 14 Patient Experience/Clinical Outcome Assessment (COA) surveys, 6 Quality of Life (QoL) assessments and are willing to allow serum concentrations of Evusheld to be drawn 9 times, 3 SARS-CoV-2 Receptor Binding Domain-Immunoglobulin G (RBD-IgG) tests, and T-cell assay to be drawn once. In the event of a symptomatic break-thru SARS-CoV-2 positive infection by SARS-COV-2 Ribonucleic Acid (RNA) by Reverse Transcription Polymerase Chain Reaction (RT-PCR) test, the patient will have an additional Evusheld serum concentration, SARS-CoV-2 RBD-IgG antibody level and T-cell assay obtained in a temporally related manner. The program requires treatment with Evusheld 600 mg IM or IV.

DETAILED DESCRIPTION:
The primary objective is to quantify the serum concentration of Evusheld (AZD7442) at 1, 2, 3, 4, 5, 6, 7, 9 or 12-months post-baseline in all qualified cancer patients treated with a single-dose of Evusheld 600 mg IM or IV at baseline.

The secondary objectives of the study are as follows:

* Compare the incidence of symptomatic Sudden Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection including SARS-CoV-2 related hospitalization and/or SARS-CoV-2 related death between solid tumor and hematologic malignancy patients.
* Compare of the incidence of symptomatic SARS-CoV-2 infection including SARS-CoV-2 related hospitalization and/or SARS-CoV-2 related death between patients treated with chemotherapy only, immunotherapy only, targeted therapy only or other/combination therapy only over 12 months post-baseline.
* Compare the serum concentration of Evusheld at 1, 2, 3, 4, 5, 6, 7, 9 and 12-months post-baseline between solid tumor and hematologic malignancy patients.
* Compare the serum concentration of Evusheld at 1, 2, 3, 4, 5, 6, 7, 9 and 12-months post-baseline between patients treated with chemotherapy only, immunotherapy only, targeted therapy only or other/combination therapy only.
* Compare of the incidence of symptomatic SARS-CoV-2 infection including SARS-CoV-2 related hospitalization and/or SARS-CoV-2 related death to the levels of serum concentration of Evusheld at 1, 2, 3, 4, 5, 6, 7, 9 and 12-months post-baseline in all patients.
* Compare the incidence of severe SARS-CoV-2 (pneumonia or hypoxemia and World Health Organization (WHO) score of ≥5) based on the TACKLE study definition between solid tumor and hematologic malignancy patients.
* Compare the incidence of severe SARS-CoV-2 (pneumonia or hypoxemia, and WHO score of ≥5) based on the TACKLE study definition death between patients treated with chemotherapy only, immunotherapy only, targeted therapy only or other/combination therapy only over 12 months post-baseline.
* Compare the incidence of severe SARS-CoV-2 (pneumonia or hypoxemia, and WHO score of ≥5) based on the TACKLE study definition to the levels of serum concentration of Evusheld at 1, 2, 3, 4, 5, 6, 7, 9 and 12-months post-baseline in all patients.
* Compare time to first event e.g., SARS-COV-2 RNA by Reverse Transcription Polymerase Chain Reaction (RT-PCR) positivity, symptomatic SARS-CoV-2 infection, hospitalization, and/or death between all four strata
* Compare Quality-of-Life metrics in all cancer patients, as measured by change from baseline to days 2, 90, 180, 270, and 360 post-baseline, and then compare the same Quality-of-Life metrics at each timepoint between each of the four strata
* Assess patient safety and adverse events including medically attended visits, Emergency Room/Urgent Care/Telehealth visits using Patient Experience/Clinical Outcome Assessment (COA) survey data for patients in each of the four strata
* Evaluate whether solid tumor or hematologic malignancy patients have a greater incidence of Evusheld-related side effects
* Assess the use of Machine Learning to predict the incidence of SARS-CoV-2 infection at days 30, 60, 90, 120, 150, 180, 210, 270 and 360 post-baseline in all cancer patients based on serum Evusheld concentration levels 3.3.3 Exploratory Objectives:
* Virologic surveillance to detect all SARS-CoV-2 variants occurring during the study in patients that test positive for SARS-CoV-2 by SARS-COV-2 RNA by Reverse Transcription Polymerase Chain Reaction (RT-PCR) testing
* Detection of potential new variants identified by positive SARS-COV-2 RNA by RT-PCR testing

ELIGIBILITY:
Inclusion Criteria:

* Male or Female gender at birth
* Age at least 18 years
* Women who are not pregnant, not breast feeding and of child bearing potential using contraception prior to enrollment in the study. Women of child bearing potential must agree to continued use of contraception throughout the 12 months of study participation.
* It is preferable that a patient has access to a "smartphone" or tablet or laptop or desktop computer and/or an email address
* In the event that a patient does not have access to any of the above, the patient may complete all follow-up surveys via the study's Call Center or in written form in the offices of the Principal Investigator as specified in the protocol
* Documented diagnosis of either hematologic malignancy or solid tumor as identified by standard ICD-10 diagnostic category
* Patients may be included with any ONE of the following criteria:
* On active treatment for solid tumor or hematologic malignancies. This can include: high-dose corticosteroids (i.e., ≥20 mg prednisone or equivalent per day when administered for ≥2 weeks), as well as any FDA-approved alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive, tumor-necrosis (TNF) blockers, and other biologic agents that are immunosuppressive or immunomodulatory (e.g., B-cell depleting agents) or any combination of these agents
* Hematologic malignancy patients can also be included if he/she is up to 12 months post-treatment and either in remission, stable or progressing as determined by the Investigator
* Solid tumor patients can also be included if he/she is up to 6 months post-treatment
* Received chimeric antigen receptor (CAR-T) or hematopoietic stem cell transplant (within 1 year of transplantation or taking immunosuppression therapy)
* Cancer is progressing as determined by the Investigator
* Treatment must have been initiated ≤12 months prior to baseline for all patients,
* Concomitant radiation therapy is permitted but cannot be the sole therapy
* Have been vaccinated with one or more doses of Janssen, Moderna or Pfizer COVID-19 vaccine
* If having been previously diagnosed with SARS-CoV-2 infection, the diagnosis has to be at least 90 days prior to study randomization. If previously diagnosed, previous treatment with Ivermectin or hydroxychloroquine is acceptable.
* Have a negative SARS-CoV-2 antigen rapid test performed in the office at screening
* Patient willing to receive treatment with AZD7442 600 mg IM or IV
* Patient willing to complete baseline and 13 post-enrollment Patient Experience/Clinical Outcome Assessment surveys.
* Patient willing to complete baseline and 5 QoL assessments
* Patient willing to have blood drawn for serum concentration of AZD7442 9 times post-baseline and repeated if patient becomes COVID-19 positive
* Patient willing to have blood drawn for T-cell assay at day 30 post-baseline and repeated if patient becomes SARS-COV-2 RNA by RT-PCR positive
* Patient willing to have RBD-IgG drawn at baseline, days 90 and 180 post-baseline and repeated if patient becomes SARS-COV-2 RNA by RT-PCR positive
* Patient willing to signed Informed Consent Form
* Patient willing to sign Authorization for Release of Health Information (including treating physicians' or other medical personnel's records, medication prescriber records, pharmacy records and medical insurance claims)

Exclusion Criteria:

* Women who are pregnant, breast feeding or of child bearing potential and not using contraception
* Absence of a qualifying type of cancer as defined by standard ICD-10 diagnostic criteria
* Treatment initiated >12 months prior to baseline or were not on active therapy ≤12 months prior to enrollment with FDA approved oral, intramuscular and/or intravenous chemotherapy, immunotherapy, targeted therapy, other therapy or any combination of these agents
* Patient receiving only radiation therapy
* Patient with an ECOG performance status of 2 or higher
* Patient with an expected cancer survival of less than 12 months by disease category
* Patient receiving adjuvant endocrine therapy as their only form of therapy for early-stage breast cancer
* Solid tumor patients more than 6 months post treatment and their cancer is considered to be stable or in remission as determined by the Investigator
* AZD7442 IM administration at any time prior to day of enrollment
* AZD7442 IM or IV administration on the same day as the patient receives any IV or IM cancer treatment
* Have a positive test for SARS-CoV-2 antigen performed by either Rapid Test or SARS-CoV-2 RNA by RT-PCR (Polymerase Chain Reaction) less than 90 days prior to enrollment
* Patient with a prior (within 90 days), current, or planned use of any of COVID-19 convalescent plasma, other monoclonal antibodies against SARS-CoV-2 or any other EUA approved SARS-CoV-2 treatment
* Patient with fever >100.0 F, and/or cough, chills, loss of smell or taste or shortness of breath or any other signs or symptoms consistent with COVID-19 within 5 days prior to enrollment
* Patient who has any known active acute respiratory infection
* Patient who has persistent (refractory to treatment for ≥14 days) bacterial or fungal infection
* Patient who has a past SARS-CoV-2 infection within 90 days prior to randomization
* Patient who has received vaccination with any dose of Janssen, Pfizer or Moderna COVID-19 vaccine less than 14 days prior to baseline for this study
* Planned use of any investigational, authorized, or approved vaccine for COVID-19 less than 14 days prior to administration of AZD7442 600 mg IM or IV
* Patient who is unwilling to have SARS-CoV-2 RBD-IgG antibody levels drawn at least 3 times
* Patient who is unwilling to receive treatment with IM or IV AZD7442
* Patient who is unwilling to complete baseline and up to 13 follow-up Experience/Clinical Outcome Assessment (COA) surveys.
* Patient who is unwilling to complete baseline and up to 5 QoL assessments
* Patient who is unwilling to have blood drawn for AZD7442 serum concentration at least 9 times
* Patient who is unwilling to have blood drawn at least once for T-cell assay
* Patient whose native language is not English and does not have a person who can translate the regulatory documents, surveys and QoL assessments.
* Patient who is unable to provide Informed Consent or Authorization for Release of Health Information due to mental illness that requires a Legally Authorized Representative.
* Patient who is legally blind and does not have a witness/caregiver who has agreed to assist the patient in his/her participation in the study.
* Patient with a history of a severe allergic reaction (i.e., anaphylaxis) to any of the components of AZD7442
* Patient with a history of severe allergic reaction (hypersensitivity) to any SARS-COV-2 vaccination, Polyethylene Glycol (PEG) or Polysorbate 80
* Patient who is illiterate and does not have a witness/caregiver who has agreed to assist the patient in his/her participation in the study.
* Patient who is participating in an interventional trial for prophylaxis or treatment of SARS-CoV-2

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
AZD7442 Serum Concentration | 12 months
  The study's primary endpoint will assess AZD7442 serum concentration collected on days 30, 60, 90, 120 150, 180, 210, 270, and 360 post-baseline in all patients.

SECONDARY OUTCOMES:
Cancer Group and Treatment Group Comparison | 12 months
  * Serum AZD7442 concentrations at 1, 2, 3, 4, 5, 6, 7, 9 and 12-months post-baseline compared between solid tumor and hematologic malignancy patients.
  * Serum AZD7442 concentrations at 1, 2, 3, 4, 5, 6, 7, 9 and 12-months post-baseline compared between patients treated with chemotherapy only, immune-therapy only, targeted therapy only or other/combination therapy only.
SARS-CoV-2 Infection | 12 months
  * Incidence of symptomatic SARS-CoV-2 infections including but not limited to those with SARS-CoV-2 related hospitalization and/or SARS-CoV-2 related death compared between solid tumor and hematologic malignancy patients.
  * Incidence of symptomatic SARS-CoV-2 infection including but not limited to SARS-CoV-2 related hospitalization and/or SARS-CoV-2 related death compared between patients treated with chemotherapy only, immunotherapy only, targeted therapy only or other/combination therapy only over 12 months post-baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Boccia, MD, Principal Investigator — Center for Cancer and Blood Disorders
Locations (40):
- United States (40):
  - Compassionate Cancer Care Medical Group, Corona, California
  - Compassionate Care Medical Group, Fountain Valley, California
  - Ventura County Hematology Oncology, Oxnard, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - Cancer Center of Southern California, Santa Monica, California
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - South Florida Cancer Care, Margate, Florida
  - Florida Cancer Affiliates-Ocala, Ocala, Florida
  - Mid-Florida Hematology Oncology Center, Orange City, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Mary Bird Perkins, Baton Rouge, Louisiana
  - Maryland Oncology Hematology, Annapolis, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Maryland Oncology Hematology, Bethesda, Maryland
  - Maryland Oncology Hematology, Brandywine, Maryland
  - Maryland Oncology Hematology, Columbia, Maryland
  - Maryland Oncology Hematology, Lanham, Maryland
  - Maryland Oncology Hematology, Rockville, Maryland
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Health Partners Institute-MMORC, Saint Louis Park, Minnesota
  - Oncology Hematology Associates, Springfield, Missouri
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Minniti Center for Oncology and Hematology, Mickleton, New Jersey
  - Southeastern Medical Oncology Center, Jacksonville, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - Alliance Cancer Specialists, Bensalem, Pennsylvania
  - Consultants in Medical Oncology Hematology, Broomall, Pennsylvania
  - Pennsylvania Cancer Specialists and Research Institute, Gettysburg, Pennsylvania
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - Alliance Cancer Specialists, Langhorne, Pennsylvania
  - Alliance Cancer Specialists, Philadelphia, Pennsylvania
  - Alliance Cancer Specialists, Sellersville, Pennsylvania
  - Alliance Cancer Specialists, Wynnewood, Pennsylvania
  - Tidelands Health Oncology, Murrells Inlet, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Summit Cancer Centers, Spokane Valley, Washington